CLINICAL TRIAL: NCT02268240
Title: Care for Post-Concussive Symptoms
Acronym: CARE4PCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: University of Washington (Other)
Responsible Party: Principal Investigator, Fred Rivara, Seattle Children's Guild Endowed Chair in Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RS_CARE4PCS
Record Dates: First submitted 2014-10-10; First posted 2014-10-20 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Stepped Care
  Interventions: Behavioral: Stepped Care
- Control (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Stepped Care — Intervention will include : 1) care management; 2) cognitive-behavioral therapy (CBT); 3) psychiatric medication consultation in addition too receiving standard care through their medical team. Care management will include initial consultation to determine participants' and families' concerns and areas of difficulty, followed by brief interventions to connect them with care providers as needed . If participants do not show adequate symptom reduction, they will be engaged in structured CBT. CBT will be delivered in 4 to 12 structured sessions, each ranging from 30-60 minutes in length. Psychiatric medication consultation will be offered on an as-needed basis for participants not adequately responding to prior stepped care interventions. MD providers with expertise in psychopharmacological treatment of youth will provide consultation for participants' primary care provider regarding the prescription of psychiatric medications.
  Arms: Experimental

SUMMARY:
The proposed study is a pilot randomized trial of a stepped collaborative care intervention designed to decrease post-concussive symptoms and improve post-injury functioning among sports-injured youth aged 11-17. Participants with persistent post-concussive symptoms (symptoms persisting at least two months post-injury) will be recruited from Seattle Children's Hospital departments of sports medicine and rehabilitation medicine. Consent and assent will be obtained in-person. Participants will be randomized to receive either the stepped collaborative care intervention, or treatment-as-usual. Participants will be assessed on a range of symptoms and areas of functioning at four time points: 0 months, 1 month, 3 months, and 6 months after enrollment. The primary hypothesis is that the intervention group athletes, when compared to usual care control group athletes, will demonstrate clinically and statistically significant reductions in postconcussive, anxiety, and depressive symptoms over the course of the 6-month study. Secondary analyses will assess the impact of the intervention on functional impairment including missed school days and other academic outcomes. Exploratory analyses will examine MRI findings that are characteristic of postconcussive neuropathology, if available in medical record, as predictors of treatment responses.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 11 and 18
* Have sustained a head impact during sports participation
* Have incurred an onset or increase of at least three post-concussive symptoms following head impact
* Have increased post-concussive symptoms following head impact have continued for at least 4 weeks
* Live with their parents or legal guardians
* Live within commuting distance of Seattle Children's Hospital
* Willing to participate in assessment and treatment
* Have at least one parent/caregiver willing to participate in assessment and treatment

Exclusion Criteria:

* Meet Diagnostic and Statistical Manual of Mental Disorders (DSM - V) criteria for a psychotic disorder or bipolar disorder
* Active suicidality
* Substance dependence

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in Concussion Symptoms | At enrollment, 1 month, 3 months, and 6 months
  Health Behavior Inventory Assessment
Change in Depressive Symptoms | At enrollment, 1 month, 3 months, and 6 months
  PHQ-9
Change in Anxiety Symptoms | At enrollment, 1 month, 3 months, and 6 months
  PROMIS A-8
Change in Quality of Life | At enrollment, 1 month, 3 months, and 6 months
  PedsQL

SECONDARY OUTCOMES:
Change in School Functioning | At enrollment, 1 month, 3 months, and 6 months
  Attendance and Grades
Change in Family Functioning | At enrollment, 1 month, 3 months, and 6 months
  FAD-GF
Change in Parent Anxiety Symptoms | At enrollment, 1 month, 3 months, and 6 months
  PROMIS A-8
Change in Parent Depressive Symptoms | At enrollment, 1 month, 3 months, and 6 months
  PHQ-9
Change in ImPACT Assessment | At enrollment and 6 months
  ImPACT test scores
NIH Toolbox - Dimensional Card Sort Test | At enrollment and 6 months
  Dimensional Card Sort Test scores
Change in NIH Toolbox - Picture Memory Sequence Test | At enrollment and 6 months
  Picture Memory Sequence test scores
Change in King-Devick Test | at enrollment and 6 months
  King-Devick Test scores

CONTACTS AND LOCATIONS:
Overall Officials: Frederick P Rivara, MD, MPH, Principal Investigator — Seattle Childrens Hospital
Locations (1):
- Seattle Childrens Hospital, Seattle, Washington, United States

REFERENCES:
- [Derived] McCarty CA, Zatzick D, Stein E, Wang J, Hilt R, Rivara FP; Seattle Sports Concussion Research Collaborative. Collaborative Care for Adolescents With Persistent Postconcussive Symptoms: A Randomized Trial. Pediatrics. 2016 Oct;138(4):e20160459. doi: 10.1542/peds.2016-0459. Epub 2016 Sep 13. PMID 27624513